CLINICAL TRIAL: NCT00404118
Title: Senior Coordinated Referral (SCORE) Study
Brief Title: Senior Coordinated Referral Study
Acronym: SCORE
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IAD 06-036
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Aged
Keywords: long-term care; satisfaction; cost
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Long-term care (LTC) can be defined as the range of institutional and home and community-based services that support individuals needing chronic care. The defining values of LTC in the VA include caring for patients in the "least restrictive environment consistent with meeting a patient's needs". VA faces an increasing demand for these services with the growing number of veterans 85 years and older, those most in need of LTC. Yet in fiscal year 2007, 87% of the 3.5 billion total VA dollars spent on LTC went to institutional care rather than the less restrictive Home and Community Based Services (HCBS). VA Central Office has formally committed to tripling the proportion of LTC that is HCBS between 1999 and 2011.

Study Objectives: (1) Develop and test measures of patient/caregiver and provider satisfaction. (2) Develop and test measures of process and cost of the LTC referrals.

Methods: Three VAMCs in VISN 11 are the study setting. This study was conducted from October 2007-June 2010 and utilized a variety of data sources throughout this timeframe. Data sources included: the Geriatric Extended Care form, telephone and in-person interviews, online and paper surveys, Extended Care Screening Committee meeting minutes, and technical reports from the Health Economics Resource Center.

Status: Complete.

DETAILED DESCRIPTION:
Long-term care (LTC) can be defined as the range of institutional and home and community-based services that support individuals needing chronic care. The defining values of LTC in the VA include caring for patients in the "least restrictive environment consistent with meeting a patient's needs". VA faces an increasing demand for these services with the number of veterans 85 years and older, those most in need of LTC. Yet in fiscal year 2007, 87% of the 3.5 billion total VA dollars spent on LTC went to institutional care rather than the less restrictive HCBS. VA Central Office has formally committed to tripling the proportion of LTC that is HCBS between 1999 and 2011.

Findings from our team's study, Assessing Practice Variation in LTC Referrals (IIR 02-228, 2006), evaluated the LTC referral process from the perspective of the referring staff, administrators, and veterans and their families. We found that the referral process is frequently unstandardized, inefficient, and not supportive of referrals to home and community-based services. VAMCs across the country have varying ways of providing LTC referrals and some look promising. Measures of the outcomes for evaluating these systems are available with the exception of two important outcomes, satisfaction with the referral and its process and cost. The goal of this study is to develop the cost and process and satisfaction measures so that such an evaluation can be conducted.

Study Objectives: (1) Develop and test measures of patient/caregiver and provider satisfaction. (2) Develop and test measures of process and cost of the referrals. The long term objective of our research is to identify and implement models of LTC referral with the best outcomes.

Methods: Three VAMCs in VISN 11 with 3 different methods of LTC referral are the study setting. This study was conducted from October 2007-June 2010 and utilized a variety of data sources throughout this timeframe. Data sources include: the Geriatric Extended Care (GEC) form, telephone and in-person interviews, online and paper surveys, Extended Care Screening Committee meeting minutes, and technical reports from the Health Economics Resource Center (HERC). The GEC forms provided recruitment information for Veterans, caregivers, social workers and nurses in both the cost and satisfaction portions of the study and were randomly pulled by the Clinical Application Coordinators at each site. Recruitment information for VA and non-VA long term care (LTC) coordinators was supplied by Site Investigators. The cost portion of the study also utilized the Extended Care Screening Committee meeting minutes and salary information for VHA employees from the HERC technical report.

Site Investigators facilitated completion of the paper surveys by attending department meetings, and coordinated in-person interviews with providers interested in participating in the study. For all telephone interviews, participants received an introduction to the study through the mail or email. Veterans and caregivers were mailed information while VA social workers, nurses, physicians and LTC coordinators were contacted via email. Potential participants then received a telephone call from a Research Assistant who further explained the study and inquired about his/her interest in participation. For the satisfaction online survey, providers were able to complete the survey after receiving the email introduction.

Status: Complete.

ELIGIBILITY:
Inclusion Criteria:

Veteran with completed Geriatrics and Extended Care Referral Form in data base at study site

Exclusion Criteria:

Inability to complete telephone interview

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients for whom a Geriatric and Extended Long-Term Care referral form was completed. For each of these patient's his/her family caregiver, provider making the referral, and long-term care program coordinator is also included.
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2007-09-25 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Development of Long-Term Care Satisfaction and Cost Measures | 09/25/2007-06/30/2010

CONTACTS AND LOCATIONS:
Overall Officials: Sheri Reder, PhD MSPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (4):
- United States (4):
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Battle Creek VA Medical Center, Battle Creek, MI, Battle Creek, Michigan
  - John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington